CLINICAL TRIAL: NCT07010120
Title: A Prospective, Single-arm Clinical Study of Immune-targeted Therapy Combined With Lysogenic HSV Virus for the Neoadjuvant Treatment of Surgically Resectable Head and Neck Squamous Carcinoma
Brief Title: A Clinical Trial of Neoadjuvant Targeted Therapy, Immunotherapy, and Lysogenic HSV-Based Virotherapy in Resectable Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024--2497
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: HNSCC; Lysogenic HSV Virus; Neoadjuvant Therapy; Immunotherapy; Targeted Therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — tislelizumab; Immunotherapy; Afatinib; Biological Factors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): 1. Tislelizumab administration on days 1 and 22, and afatinib continuous administration from days 1 to 42
  2. Lysosomal HSV virus injection (divided into a dose-escalation phase and a dose-expansion phase; in the dose-escalation phase, Group 1 took 106 pfu/mL and Group 2 took 108 pfu/mL, and in the dose-expansion phase the dose of lysosomal HSV virus with the highest MPR of the escalation phase was taken.) .. The dose of intralymph node injection of lysosomal HSV virus in patients was determined according to the size of metastatic lymph nodes, (diameter less than or equal to 1.5 cm, maximum 1 mL; diameter 1.5-2.5 cm, maximum 2 mL; diameter greater than 2.5 cm, maximum 4 mL). Two injections were given per patient, with each dose separated by 2 weeks.
  3. Standard of care surgery
  Interventions: Drug: Tislelizumab; Drug: Afatinib; Biological: Lysogenic HSV virus.

INTERVENTIONS:
Drug: Tislelizumab — 200mg IV Q3W
  Other Names: Immunotherapy
Drug: Afatinib — 30mg PO QD
  Other Names: Targeted therapy
Biological: Lysogenic HSV virus. — Lysosomal HSV virus injection (divided into a dose-escalation phase and a dose-expansion phase; in the dose-escalation phase, Group 1 took 106 pfu/mL and Group 2 took 108 pfu/mL, and in the dose-expansion phase the dose of lysosomal HSV virus with the highest MPR of the escalation phase was taken.) .. The dose of intralymph node injection of lysosomal HSV virus in patients was determined according to the size of metastatic lymph nodes, (diameter less than or equal to 1.5 cm, maximum 1 mL; diameter 1.5-2.5 cm, maximum 2 mL; diameter greater than 2.5 cm, maximum 4 mL). Two injections were given per patient, with each dose separated by 2 weeks.
  Other Names: Biological agent

SUMMARY:
Evaluation of the safety and tolerability of immune-targeted therapy combined with neoadjuvant therapy with lysogenic HSV virus for patients with surgically resectable squamous carcinoma of the head and neck.

DETAILED DESCRIPTION:
Head and Neck Squamous Cell Carcinoma (HNSCC) is one of the most common malignant tumors in the head and neck region. Globally, both its incidence and mortality rates have shown a significant upward trend, posing a serious threat to the life and health of patients.

Although surgical resection is the main treatment approach for resectable HNSCC, a considerable number of patients still face a high risk of local recurrence and distant metastasis after surgery, which are the key factors contributing to poor prognosis.

In recent years, immune-targeted therapy has emerged in the field of malignant tumor treatment and demonstrated unique treatment advantages and potential. It can specifically act on relevant targets of tumor cells, precisely regulate the body's immune system, and effectively enhance the body's immune response to tumor cells, thereby inhibiting the malignant biological behaviors of tumor cells such as growth, proliferation, and metastasis. Oncolytic herpes simplex virus (HSV) has the ability to specifically replicate within tumor cells and lyse them. Meanwhile, it can also induce a strong anti-tumor immune response in the body and has broad application prospects in tumor treatment.

Based on the above situation, this study innovatively proposes to combine immune-targeted therapy with oncolytic HSV virus for the neoadjuvant treatment of resectable HNSCC. The aim is to fully utilize the synergistic effect of the two treatment modalities, minimize the tumor volume to the greatest extent, reduce the tumor stage, improve the surgical resection rate and radicality, decrease the risks of postoperative recurrence and metastasis, and ultimately improve the quality of life and prognosis of patients. By conducting this prospective, single-arm clinical study, it is expected to provide a more efficient, safe, and innovative treatment strategy and clinical practice basis for the treatment of resectable HNSCC.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 and ≤70 years old, regardless of gender;

Patients with head and neck squamous carcinoma who are pathologically confirmed and fulfill the following conditions:

Patients with locally advanced head and neck squamous carcinoma (excluding nasopharyngeal, salivary gland and thyroid malignant tumors) who are initially diagnosed and have no distant metastasis;

Non oropharyngeal HNSCC carcinoma and HPV-negative oropharyngeal carcinoma, stages III, IVA and IVB; HPV-positive oropharyngeal cancers, stages II and III; HPV status of oropharyngeal cancer will be determined by p16 immunohistochemistry.

Treatable by surgical resection as evaluated by head and neck surgery; Definite lymph node metastasis and lymph node stage is not N0 or Nx. An Eastern Cooperative Oncology Group (ECOG) physical status score of 0 to 1;

Have adequate organ and bone marrow function as defined below:

Subjects voluntarily enrolled in the study, signed an informed consent form, and were able to comply with the visits and related procedures specified in the protocol.

Exclusion Criteria:

Lymph node staging of N0 or Nx status; History of other malignancies (except history of cured and non-recurrent basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, cervical cancer in situ, intramucosal carcinoma of the gastrointestinal tract, and other malignancies considered by the investigator to be eligible for enrollment); Any active autoimmune disease or history of autoimmune disease including, but not limited to, immune-related neurological disorders, multiple sclerosis, autoimmune (demyelinating) neuropathies, Guillain-Barre Syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease including Crohn's disease and ulcerative colitis, autoimmune hepatitis, toxic epidermal Necrolytic Elastosis (TEN) or Stevens-Johnson Syndrome (except for type I diabetes on stabilized doses of insulin); A history of anaphylaxis, severe drug allergy, known allergy to any component of a large protein preparation, PD-1 monoclonal antibody injection, or afatinib prescription (Note: severe allergy is defined as resulting in hospitalization);

Received any of the following treatments:

Patients with prior use of PD-1 antibody, PD-L1 antibody, CTLA-4 antibody, EGFR antibody, or EGFR-TKI; Patients who have received an anti-tumor vaccine; Use of any active vaccine against infectious diseases (e.g., influenza vaccine, varicella vaccine, etc.) within 4 weeks prior to the first dose or scheduled to be used during the study period; Major surgery or severe trauma within 4 weeks prior to the first dose of study drug; Inhaled or topical steroids and adrenal hormones (>10 mg/day of prednisone) are permitted as an alternative therapy for patients requiring systemic therapy with corticosteroids (>10 mg/day of prednisone) or other immunosuppressive agents within 14 days prior to administration of study drug; Those with serious medical conditions such as abnormal class II or higher cardiac function (NYHA criteria), ischemic heart disease (e.g., myocardial infarction or angina pectoris), clinically significant supraventricular or ventricular arrhythmia with echocardiographic ejection fraction <50%; QTc interval, >450 msec in men and >470 msec in women; and an abnormal electrocardiogram that, in the opinion of the investigator, poses an experimental drug There is an additional risk; Subjects with a known history of interstitial pneumonia, history of non-infectious pneumonia, or a high suspicion of interstitial pneumonia; or subjects who may interfere with the detection or management of suspected drug-related pulmonary toxicity; subjects with a prior history of pharmacogenetic or radiologic non-infectious pneumonia that is asymptomatic are permitted to enroll in the study; subjects with active tuberculosis, or with a history of prior tuberculosis infection that has not been controlled with treatment; Patients with hyperthyroidism and patients with organic thyroid disease are not eligible for enrollment; hypothyroidism treated with a stable dose of thyroid replacement hormone is eligible for enrollment, and hypothyroidism that can be controlled with thyroid replacement hormone treatment is eligible for enrollment (control or not will be confirmed by the investigator and/or the endocrinology department); Presence of an active infection, or fever of unknown origin during screening, 48 h prior to the first dose, or use of systemic antibiotics within 1 week prior to signing informed consent; Presence of active hepatitis B (HBV DNA ≥ 2000 IU/ml or 104 copies/ml) or hepatitis C (hepatitis C antibody positive with HCV RNA above the lower limit of detection of the analytical method), or known history of positive human immunodeficiency virus (HIV) test or known acquired immunodeficiency syndrome (AIDS); A previous history of a definite neurologic or psychiatric disorder, such as epilepsy or dementia; a definite history of substance abuse or a history of alcohol abuse within 3 months; women who are pregnant or breastfeeding; subjects (and their partners) who have plans to have children, have sex without contraception, or are unwilling to use adequate contraception (e.g., use of condoms, contraceptive rings, or partner sterilization) during the screening period to 3 months after the end of their study; Received any investigational drug within 4 weeks prior to the first dose of study drug or concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or an interventional clinical study follow-up; In the judgment of the investigator, the subject may have other factors affecting this study that would prevent completion of the trial medication and follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 29 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity (DLT) Incidence. | Intraoperative.
  Dose-Limiting Toxicity (DLT) is the maximum safe dose of radiotherapy that a patient can tolerate in an experiment.

SECONDARY OUTCOMES:
Major Pathologic Response | Intraoperative.
  c Response (MPR) was defined as fewer than 10% viable tumor cells.
Pathologic Complete Response | Intraoperative.
  Pathologic Complete Response (pCR) was defined as the absence of viable tumor cells.
Objective Response Rate | Up to 8 weeks
  Objective Response Rate (ORR) was defined as the percentage of participants with a best overall response of CR or PR using RECIST Criteria
Adverse events | Up to 12 weeks
  Adverse events were defined as the number of participants with adverse events using CTCAE Criteria or with an unplanned surgery delay.
Disease-free Survival | 1 year
  Disease-free Survival (DFS) was defined as the time from the administration of the first dose to first disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- Department of Radiation Oncology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Pulte D, Brenner H. Changes in survival in head and neck cancers in the late 20th and early 21st century: a period analysis. Oncologist. 2010;15(9):994-1001. doi: 10.1634/theoncologist.2009-0289. Epub 2010 Aug 26. PMID 20798198
- [Background] Denaro N, Merlano MC, Russi EG. Follow-up in Head and Neck Cancer: Do More Does It Mean Do Better? A Systematic Review and Our Proposal Based on Our Experience. Clin Exp Otorhinolaryngol. 2016 Dec;9(4):287-297. doi: 10.21053/ceo.2015.00976. Epub 2016 Jun 25. PMID 27337948
- [Background] Harari PM. Promising new advances in head and neck radiotherapy. Ann Oncol. 2005;16 Suppl 6:vi13-vi19. doi: 10.1093/annonc/mdi453. PMID 15987991
- [Background] Haddad R, O'Neill A, Rabinowits G, Tishler R, Khuri F, Adkins D, Clark J, Sarlis N, Lorch J, Beitler JJ, Limaye S, Riley S, Posner M. Induction chemotherapy followed by concurrent chemoradiotherapy (sequential chemoradiotherapy) versus concurrent chemoradiotherapy alone in locally advanced head and neck cancer (PARADIGM): a randomised phase 3 trial. Lancet Oncol. 2013 Mar;14(3):257-64. doi: 10.1016/S1470-2045(13)70011-1. Epub 2013 Feb 13. PMID 23414589
- [Background] Machiels JP, Haddad RI, Fayette J, Licitra LF, Tahara M, Vermorken JB, Clement PM, Gauler T, Cupissol D, Grau JJ, Guigay J, Caponigro F, de Castro G Jr, de Souza Viana L, Keilholz U, Del Campo JM, Cong XJ, Ehrnrooth E, Cohen EE; LUX-H&N 1 investigators. Afatinib versus methotrexate as second-line treatment in patients with recurrent or metastatic squamous-cell carcinoma of the head and neck progressing on or after platinum-based therapy (LUX-Head & Neck 1): an open-label, randomised phase 3 trial. Lancet Oncol. 2015 May;16(5):583-94. doi: 10.1016/S1470-2045(15)70124-5. Epub 2015 Apr 16. PMID 25892145